CLINICAL TRIAL: NCT04806737
Title: A Phase IIa, Double-blind, Randomised, Placebo-controlled Study on the Efficacy and Tolerability of a 14-day Treatment With Teriflunomide vs. Placebo in Subjects With Coeliac Disease Undergoing a 3-day Gluten Challenge
Brief Title: Teriflunomide vs. Placebo During Gluten Challenge in Celiac Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Knut E. A. Lundin, Professor, M.D., PhD., Consultant gastroenterologist, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-002307-18
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Celiac Disease
Keywords: Immunotherapy; Gluten challenge; Teriflunomide
MeSH Terms: conditions — Celiac Disease | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMP (Active Comparator): Teriflunomide 14 mg tablets, first 7 days 5 tablets once pr day, thereafter 1 pr day for another 6 days.
  Interventions: Drug: Teriflunomide Oral Tablet
- Placebo (Placebo Comparator): Sham tablets
  Interventions: Drug: Teriflunomide Oral Tablet

INTERVENTIONS:
Drug: Teriflunomide Oral Tablet — The study will be conducted with two treatment groups in the form of a 2:1 parallel group comparison and will serve to compare oral treatment with 14 mg/d teriflunomide vs. placebo in subjects with well-controlled coeliac disease undergoing gluten challenge. The screening period will be up to 8 weeks, followed by a 7-day run-in treatment period with a loading dose of teriflunomide followed by a 6 day therapeutic maintenance dose, an initial 4-week treatment-free follow-up period and a 6 month closing follow-up.
  Other Names: Gluten challenge

SUMMARY:
The investigators will see if the drug teriflunomide (which is in use in other immune disorder (multiple sclerosis)) can inhibit the immune activation in celiac disease patients during a 3 day gluten challenge. This will be measured in a blood sample.

DETAILED DESCRIPTION:
This is a controlled, double-blind, randomised, singlecentre, placebo-controlled, phase IIa proof-of-concept study on effects of the drug on activation and efflux of gluten specific T cells using HLA-DQ:gluten tetramers. The study will be conducted with two treatment groups in the form of a 2:1 parallel group comparison and will serve to compare oral treatment with 14 mg/d teriflunomide vs. placebo in subjects with well-controlled coeliac disease undergoing gluten challenge. The screening period will be up to 8 weeks, followed by a 7-day run-in treatment period with a loading dose of teriflunomide followed by a 6 day therapeutic maintenance dose, an initial 4-week treatment-free follow-up period and a 6 month closing follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-80
* Willingness to comply with the study procedures and having signed informed, written consent
* Previous diagnosis of coeliac disease according to established guidelines based on positive serology (Endomysium test, IgA-TG2 and/or IgGDGP) and a duodenal biopsy showing villous atrophy graded as Marsh 3
* Positive gene test for HLA-DQ2.5
* Adherence to gluten-free diet

Exclusion Criteria:

* Known intolerance to ingredients of teriflunomide or placebo tablets
* Known intolerance to gluten challenge
* Known intolerance to cholestyramine
* Duration of gluten free diet shorter than six months
* Positive serology (IgA-TG2 below upper level of normal) at screening visit
* Pregnancy or breast-feeding
* Not willing to comply with proper pregnancy control (in females)
* Concomitant medication that interferes with immune activation (e.g. steroids, calcineurin inhibitors, biological treatment for inflammatory bowel disease or other immune disorders, further list is given below)
* Any other medical condition that in the opinion of the principal investigator makes the individual unsuitable for participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Adaptive T cell activation | Blood sample on the 4th day after a 3 day gluten challenge
  Expression of CD38 on HLA-DQ:gluten tetramer positive T cells

CONTACTS AND LOCATIONS:
Overall Officials: Pål-Dag Line, MD, PhD, Study Chair — Oslo University Hoapital; Knut EA Lundin, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Dept of Gastroenterology, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No